CLINICAL TRIAL: NCT03512795
Title: Optimization of HIV-1 DNA Genotyping by High Throughput Sequencing to Document Antiretroviral Resistant Mutations
Acronym: Mutapro
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: BLOT AOI 2017
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Blood samples — An additional blood tube will be taken during the patient's follow-up blood collection.

SUMMARY:
The analysis of HIV resistance to antiretrovirals (Sanger sequencing on RNA) is difficult when the viral load is undetectable or during therapeutic breaks. In these situations, the ultra-deep sequencing (UDS) can be done on proviral DNA in order to improve characterization of archived resistant variants with may reflect past virological failures.

This study is a cross-sectional study which will require only one additional tube which can be taken during a routine check-up as part of the usual follow-up of the individuals included.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has given consent
* Adult patient
* Patient living with HIV-1
* Controlled viral load (<50 RNA copies/ml) for at least 1 year.
* At least two previous virologic failures, either :

  * Initial failure : defined as the persistence of a viral load greater than 50 copies/ml beyond 1 year, after the initiation of triple antiretroviral therapy, and without virological control (VL > 50 copies/ml) since the initiation of the very first antiretroviral treatment.
  * A rebound in HIV viral load to more than 50 copies/ml after a period of virological success, confirmed on two consecutive samples at least one month apart.
* At least 2 Sanger RNA genotypes have been done or could be done from the existing library.

Exclusion Criteria:

* Patient not affiliated to a medical insurance scheme
* Protected adult
* Pregnant, parturient or breastfeeding woman
* Discontinuation of clinical and immuno-virological follow-up for more than 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients living with HIV-1, with an undetectable viral load and a history of at least 2 virological failures in which resistance to at least two drug classes was observed
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
> Genotyping Score (GSS) comparison between HIV DNA-UDS genotyping assay obtained at inclusion and cumulative RNA-Sanger genotyping assays obtained at each virological failure during routine follow | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France